CLINICAL TRIAL: NCT06837025
Title: The Efficacy of Fascial Manipulation Compared to Stretching in the Rehabilitation of Children With Cerebral Palsy
Brief Title: Fascial Manipulation in Cerebral Palsy Rehabilitation
Acronym: CP fascia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orton Orthopaedic Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2500/511; A2500/511 (Other Grant/Funding Number: This is supported by Research Institute Orton through grants by the Ministry of Social Affairs and Health in Finland)
Record Dates: First submitted 2025-01-31; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Fascial manipulation; Flexibility; Spasticity; Walking ability; Interview study; qualitative study
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial manipulation (Active Comparator): In fascia manipulation (FM), the treatment targets the deep fascia related to muscles, including the aponeurotic and epimysial fascia. Treatment points are selected based on a thorough assessment, including the client's history, movement tests and analysis, and palpation tests. Fascia manipulation treatment affects the hyaluronan and viscosity of the muscle fascia. In the treatment of spasticity, the treatment points are in the body parts involved in spastic movement patterns. In this study, fascia manipulation is performed once a week, and the therapist provides instructions for self-exercises to the child with CP.
  The child's own physiotherapy continues at the same time.
  Interventions: Other: Fascial manipulation
- Stretching (Active Comparator): The stretches are based on the article published 2024 at University of Jyväskylä. Four sets of 45-second manual passive-static guided stretches to the pain threshold are performed for the ankle extensors, hip flexors, hip adductors, and knee flexors.
  Interventions: Other: Fascial manipulation

INTERVENTIONS:
Other: Fascial manipulation — Fascial manipulation once a week
  Other Names: 1

SUMMARY:
The purpose of the study is to investigate the potential additional benefits of a relatively new physiotherapy method, fascial manipulation, in the rehabilitation of movement difficulties or other problems caused by CP (cerebral palsy). A physiotherapist specialized in fascial manipulation specifically treats the muscle fascia, which plays a central role in the problems associated with CP. Fascial manipulation feels just like a massage but does not hurt.

The purpose of the study is to determine how physiotherapeutic rehabilitation methods should be further developed in Finland and elsewhere. Fascial manipulation was originally developed in Italy and is used to treat many musculoskeletal problems. There have been few studies on the effectiveness of fascial manipulation in the context of CP problems. It is important to obtain more research evidence, which is why conducting this study is crucial.

DETAILED DESCRIPTION:
Introduction Fascial manipulation (FM) is a manual therapy method developed by physiotherapist Luigi Stecco. It involves the treatment of deep fascia related to muscles or superficial fascia of subcutaneous tissue, which is made up of connective tissue. The goal of FM is to normalize the function of muscle-related fascia, allowing movement to return to normal and overstrained or painful structures to heal. Superficial fascial treatment is needed, for example, in the treatment of surgical scars and swelling The method has been used to treat various musculoskeletal disorders, with evidence supporting its effectiveness.

FM can be used in the rehabilitation of children with CP (cerebral palsy) to treat stiffness caused by the non-neural component of spasticity. Both neural and non-neural factors influence the abnormal movement patterns caused by spasticity in children with CP. Recent research suggests that non-neural factors are functionally more significant.

Spasticity caused by upper motor neuron damage leads to an increase in the extracellular matrix (ECM) of the muscle. The main component of the extracellular matrix is hyaluronan (HA), which facilitates internal muscle and intermuscular sliding and myofascial force transmission.

The mechanical properties of the muscle, such as stiffness and viscosity, often change with spasticity, as the increased concentration of HA associated with spasticity can increase the viscosity of the ECM and the collagen content in the muscle. This affects both active and passive movement and alters the force production and coordination between agonist and antagonist muscles. Increased resistance to active movement causes fatigue and pain. Increased ECM viscosity increases the stretch on the perimysium and the muscle spindle attached to it, sensitizing spindle activation. These non-neural peripheral factors are believed to cause muscle stiffness.

There have been few studies on the effectiveness of FM in the rehabilitation of children with CP. The limited studies and practical observations suggest that treatment targeting muscle-related fascia may be a beneficial addition to the rehabilitation of children with CP. High-quality studies on the effectiveness of FM in general musculoskeletal rehabilitation are scarce. A recent systematic review indicates that the level of evidence for FM is low to moderate. A systematic review on children with CP has recently been published.

In Finland, the rehabilitation of children with CP has largely relied on the NDT/Bobath framework, although its effectiveness has been strongly criticized in a recent meta-analysis. The need for further research is evident.

Therapists trained in NDT/Bobath use their experience, reflection, and knowledge gained from various continuing education courses in their work. The NDT-Bobath approach serves as the framework for clinical decision-making in therapy. It emphasizes the importance of the child's own activity in the development of agency.

Research Objectives The aim is that the therapy method used in the study will provide additional benefits to the rehabilitation of children with CP by enabling better movement patterns, more effective training, and more economical movement, thereby enhancing the child's/youth's functional capacity. The indication for fascia manipulation is to prevent and correct the typical functional limitations caused by CP and to enable better functional capacity.

Based on clinical observations, the acute effect of FM on the movement of children with CP is promising. The aim of this study is to investigate the acute and longer-term effects of FM using objective methods. The researchers will conduct an eight-week randomized and controlled rehabilitation intervention study with children with CP, comparing the effect of FM on walking ability and lower limb joint movements to therapy conducted according to current best rehabilitation practices. Through an interview study (with parents after the intervention), the researchers will investigate the potential added value of FM in the participant's involvement and empowerment, i.e., the ability to participate more diversely in various social activities and cope with hobbies, school, and other community activities. The assumption is that movement will be less strenuous. An interview with the child's own physiotherapist after the fascia manipulation intervention aims to identify any changes in functional capacity and therapy situations observed by the physiotherapist.

The Gross Motor Function Classification Scale (GMFCS) is used to determine the severity of the motor impairment in children with CP, describing gross motor function, i.e., movement. The classification uses levels 1-5 (Terveyskylä, Lastentalo, CP-vamma lapsella). The target group for this study are children at GMFCS level 2 (independent walking without assistive devices, often requiring orthoses, with some difficulty moving outside the home, e.g., stairs) and GMFCS level 3 (independent walking with assistive devices, such as a walker or rollator, with significant difficulty moving outside the home, often using a wheelchair outdoors).

Hypotheses:

I) Acute Effect: Compared to conventional neurological physiotherapy, fascia manipulation more effectively reduces spasticity and stiffness in the ankle and other lower limb joints and decreases co-contraction of the extensor-flexor muscles of the ankle during walking. Participants will include those in GMFCS levels 2 and 3. They rarely have differentiated movement in the ankle, so any changes will be visible in the movements of the knee and hip.

II) Longitudinal Effect: Compared to conventional neurological physiotherapy, fascia manipulation treatment better promotes the function of lower limb joints, which is reflected in an improved walking pattern (Gait Deviation Index) and positive changes in walking performance (6-minute walk test, primary outcome measure) and efficiency (oxygen consumption).

III) Improved mobility increases and eases patients' participation in various activities outside the home, such as attending school and engaging in hobbies, and transitions in these situations

Study Design and Patient Recruitment

The researchers will conduct an 8-week randomized and controlled rehabilitation intervention study, recruiting 20 children aged 7-14 years with a diagnosis of spastic CP (GMFCS levels 2-3) . The participants will be recruited from the HUS/ULS patient registry.

Sample Size and Randomization

Power calculations were performed based on the primary outcome measure (6-minute walk test). Based on clinical observations, the researchers estimate that FM increases walking speed by approximately 10% (0.05 m/s), which corresponds to an improvement of about 60 meters in the 6-minute walk test. With an effect size of 0.8, the required sample size would be 15 (power = 90% and α = 0.05), but the researchers are accounting for a 25% dropout rate and will recruit a total of 20 children with CP.

Participants will be randomized into two groups of 10: 1) fascia manipulation group (intervention group I) and 2) conventional physiotherapy group (intervention group II). Randomization will be done in blocks of four based on age, gender, GMFCS level, and baseline walking ability (6-minute test) and walking pattern (Gait Deviation Index). Once a group of four participants is formed based on registry data, they will be contacted, and both the child and the guardian will be asked about their willingness to participate in the study. If the child and guardian are willing to participate, the participants will be assigned to groups using a computer-based randomization tool, distributing 2-4 participants (considering GMFCS level, age, gender, and 6-minute walk test result) to intervention group I and intervention group II. If the child or guardian declines, a new participant will be sought using registry data (considering age, gender, and severity of CP), and their willingness to participate in the study will be asked. This process will continue until the intervention groups are formed.

The study is prepared to increase the sample size by an additional 10 (5+5) patients if necessary. The decision will be made after 20 (10+10) patients have been studied and the interventions have been carried out. If there is attrition or other issues that complicate statistical analysis, the sample size will be increased.

Intervention Group I

In Intervention Group I, children will undergo motion analysis measurements at the beginning of the study, receive one fascia manipulation treatment, and then have the measurements repeated after the treatment to assess the acute response to the therapy. The group will receive 8 FM intervention treatments (once a week) either at the child's home or at the physiotherapist's office. The therapy intervention will last about two months. After the treatments, the children will undergo motion analysis measurements again to assess the longitudinal effect of the therapy. It is noteworthy that during the fascia manipulation treatment, the regular weekly physiotherapy based on stretching will continue.

Intervention Group II

In Intervention Group II, children will undergo initial measurements, after which the physiotherapist will guide them through stretching exercises, and final measurements will be taken to assess the acute response to the stretching. During the two-month intervention, the children will receive the same therapy as before (traditional physiotherapy) and, in addition, a remotely conducted stretching program guided by the physiotherapist. Thus, the children will receive physiotherapy twice a week. This arrangement is to more reliably assess the potential added value of fascia manipulation. After the two-month intervention, the children in Intervention Group II will undergo the same motion analysis measurements as at the beginning, and then Intervention Group II will receive FM therapy eight times. The duration of the intervention is about two months.

A semi-structured interview will be conducted with the relative (parent) of the participant after the fascia manipulation intervention. A total of about 10 parents will be interviewed. The aim of the qualitative study is to document the impact of FM on the participant's daily life, schooling, social participation, and the effects on the lives of the participant's parents. The study will also interview the participant's physiotherapist (a total of about 10). The researcher will contact the interviewee to arrange a suitable time. The interview can be conducted either via Teams remote connection or face-to-face. The interview will last about 30 minutes. The interviews will be recorded if the interviewees give their consent. The recorded interviews will be transcribed anonymously, and personal data will not be linked to the anonymized data.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-14 years
* GMFCS level 2-3
* Good cooperation
* Family living in the Helsinki metropolitan area

Exclusion Criteria:

* The child has previously received fascia manipulation by a Stecco-trained therapist or other fascia treatment (if done within the last 6 months)
* Surgeries on the lower limbs (if done within the last 12 months)
* Electrical stimulation treatments (if done within the last 3 months)
* Botox treatments on the lower limbs (if done within the last 6 months)
* Reduced cognitive level
* Severe visual impairment (unable to perform the walking test)
* Other illnesses: psychological or other serious illness

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-minute walking test | From enrollment to the end of treatment at 8 weeks
  Distance covered six minutes

SECONDARY OUTCOMES:
Walking efficiency | From enrollment to the end of treatment at 8 weeks
  Efficiency determined by respiratory gas analyser.
  Walking efficiency is determined by calculating the energy cost of walking using following formula:
  Energy cost (J/kg/m) = (4.960 × respiratory exchange ratio + 16.040) × VO2 (ml/kg/min)/walking speed (m/min). The respiratory exchange ratio is calculated by dividing VO2 by VCO2. VO2 and VCO2 are the average oxygen uptake and carbon dioxide production during the last 2 minutes of the 6-min walking test respectively, relative to body weight (ml/kg/min). Mobile metabolic system Cormed K5 will be used to collect VO2 and VCO2 data.
Ankle joint hyper-resistance | From enrollment to the end of treatment at 8 weeks
  Ankle spasticity measured in an isokinetic dynamometer and electromyography.
  Ankle joint hyper-resistance is assessed using an isokinetic dynamometer (Contrex) by measuring passive joint torques at slow (10 deg/s) and fast speeds (300 deg/s). The appropriate range of motion for the foot attachment is determined during the pre-test by moving the ankle towards dorsiflexion until the passive torque reaches 10-15 Nm. This same range of motion will be used during the post-test to allow for pre-post comparison. Measurements at low speed indicate passive ankle joint stiffness, while measurements at fast speed indicate stretch hyperreflexia (or spasticity).
Gait pattern | From enrollment to the end of treatment at 8 weeks
  Gait Deviation Index measured during walking during walking by 3D motion analysis.
  A GDI (gait deviation index, scale 0-100) score of 100 indicates a gait pattern similar to the normative data, while lower scores indicate greater deviations from the normal. Every ten points is one standard deviation away from the normative mean. Vicon motion analysis system is used to collect gait data.
Interview: Parents of a child with cerebral palsy and their physiotherapist | From enrollment to the end of treatment at 8 weeks
  How does a child with cerebral palsy manage with everyday life? What observations do the parents and the child's physiotherapist make during the research intervention?

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tolvanen 2019 http://www.fascialmanipulation.com/wp-content/uploads/ATTI-2019-PDF.pdf
- [Result] Tolvanen 2018, Treatment of neurological pediatric patients in Julia Ann Day, Fascial Manipulation-Stecco -method The practitioner´s perspective, Handspring .
- [Result] Tolvanen, Lahtinen-Suopanki, 2022, Fascia Research Congress (poster), The Experiences and Benefits of Applying Fascial Manipulation® Stecco Method in Neurological Physiotherapy for Children and Adults. https://www.fasciaresearchsociety.org/docs/2022_FRC_AbstractBook.pdf
- [Result] BOBATH K, BOBATH B. THE FACILITATION OF NORMAL POSTURAL REACTIONS AND MOVEMENTS IN THE TREATMENT OF CEREBRAL PALSY. Physiotherapy. 1964 Aug;50:246-62. No abstract available. PMID 14179895
- [Result] Stecco L, Basmanjian JV, Day JA. (2004). Fascial manipulation for musculoskeletal pain (pp. 123-130). Padova: Piccin.
- [Result] Stecco A, Raghavan P: Peripheral Mechanisms Contributing to Spasticity and Implications for Treatment. Curr Phys Med Rehabil Rep. 2014;2:121-127. DOI 10.1007/s40141-014-0052-3.
- [Result] Hansen AB, Price KS, Loi EC, Buysse CA, Jaramillo TM, Pico EL, Feldman HM. Gait changes following myofascial structural integration (Rolfing) observed in 2 children with cerebral palsy. J Evid Based Complementary Altern Med. 2014 Oct;19(4):297-300. doi: 10.1177/2156587214540466. Epub 2014 Jul 2. PMID 24989994
- [Result] Pintucci M, Simis M, Imamura M, Pratelli E, Stecco A, Ozcakar L, Battistella LR. Successful treatment of rotator cuff tear using Fascial Manipulation(R) in a stroke patient. J Bodyw Mov Ther. 2017 Jul;21(3):653-657. doi: 10.1016/j.jbmt.2016.12.007. Epub 2016 Dec 22. PMID 28750980
- [Result] Faccioli S, Pagliano E, Ferrari A, Maghini C, Siani MF, Sgherri G, Cappetta G, Borelli G, Farella GM, Foscan M, Vigano M, Sghedoni S, Perazza S, Sassi S. Evidence-based management and motor rehabilitation of cerebral palsy children and adolescents: a systematic review. Front Neurol. 2023 May 25;14:1171224. doi: 10.3389/fneur.2023.1171224. eCollection 2023. PMID 37305763
- [Result] Amir A, Kim S, Stecco A, Jankowski MP, Raghavan P. Hyaluronan homeostasis and its role in pain and muscle stiffness. PM R. 2022 Dec;14(12):1490-1496. doi: 10.1002/pmrj.12771. Epub 2022 Feb 25. PMID 35077007
- [Result] Cowman MK, Schmidt TA, Raghavan P, Stecco A. Viscoelastic Properties of Hyaluronan in Physiological Conditions. F1000Res. 2015 Aug 25;4:622. doi: 10.12688/f1000research.6885.1. eCollection 2015. PMID 26594344
- [Result] Smith LR, Lee KS, Ward SR, Chambers HG, Lieber RL. Hamstring contractures in children with spastic cerebral palsy result from a stiffer extracellular matrix and increased in vivo sarcomere length. J Physiol. 2011 May 15;589(Pt 10):2625-39. doi: 10.1113/jphysiol.2010.203364. Epub 2011 Mar 21. PMID 21486759
- [Result] Menon RG, Oswald SF, Raghavan P, Regatte RR, Stecco A. T1rho-Mapping for Musculoskeletal Pain Diagnosis: Case Series of Variation of Water Bound Glycosaminoglycans Quantification before and after Fascial Manipulation(R) in Subjects with Elbow Pain. Int J Environ Res Public Health. 2020 Jan 22;17(3):708. doi: 10.3390/ijerph17030708. PMID 31979044
- [Result] Valadao P, Cenni F, Piitulainen H, Avela J, Finni T. Effects of the EXECP Intervention on Motor Function, Muscle Strength, and Joint Flexibility in Individuals with Cerebral Palsy. Med Sci Sports Exerc. 2024 Jan 1;56(1):1-12. doi: 10.1249/MSS.0000000000003273. Epub 2023 Aug 7. PMID 37565430
- [Result] Te Velde A, Morgan C, Finch-Edmondson M, McNamara L, McNamara M, Paton MCB, Stanton E, Webb A, Badawi N, Novak I. Neurodevelopmental Therapy for Cerebral Palsy: A Meta-analysis. Pediatrics. 2022 Jun 1;149(6):e2021055061. doi: 10.1542/peds.2021-055061. PMID 35607928
- [Result] Arumugam K, Harikesavan K. Effectiveness of fascial manipulation on pain and disability in musculoskeletal conditions. A systematic review. J Bodyw Mov Ther. 2021 Jan;25:230-239. doi: 10.1016/j.jbmt.2020.11.005. Epub 2020 Nov 11. PMID 33714501
- [Result] Raghavan P, Lu Y, Mirchandani M, Stecco A. Human Recombinant Hyaluronidase Injections For Upper Limb Muscle Stiffness in Individuals With Cerebral Injury: A Case Series. EBioMedicine. 2016 Jul;9:306-313. doi: 10.1016/j.ebiom.2016.05.014. Epub 2016 May 13. PMID 27333050
- [Result] Nielsen JB, Christensen MS, Farmer SF, Lorentzen J. Spastic movement disorder: should we forget hyperexcitable stretch reflexes and start talking about inappropriate prediction of sensory consequences of movement? Exp Brain Res. 2020 Aug;238(7-8):1627-1636. doi: 10.1007/s00221-020-05792-0. Epub 2020 May 7. PMID 32382862
- [Result] Stecco A, Stern R, Fantoni I, De Caro R, Stecco C. Fascial Disorders: Implications for Treatment. PM R. 2016 Feb;8(2):161-8. doi: 10.1016/j.pmrj.2015.06.006. Epub 2015 Jun 14. PMID 26079868